CLINICAL TRIAL: NCT00588003
Title: Analysis of Gene Expression Following Short Term Exposure to Neoadjuvant Endocrine Therapy in Invasive Breast Cancer
Brief Title: Gene Expression Following Short Term Exposure to Neoadjuvant Endocrine Therapy in Invasive Breast Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None
Other Study IDs: 03-153
Record Dates: First submitted 2007-12-22; First posted 2008-01-08 (Estimated); Last update posted 2015-12-24 (Estimated); Status verified 2015-12

CONDITIONS: Breast Cancer
Keywords: Breast; ANASTROZOLE
MeSH Terms: conditions — Breast Neoplasms | interventions — Anastrozole

ARMS (2):
- 1 (Experimental): This is an exploratory study utilizing micro-array technology and immunohistochemistry to test the hypothesis that changes in gene expression occur as an early event in response to endocrine therapy and that these changes can be correlated with changes in surrogate biological markers.
  Interventions: Drug: anastrozole
- 2 (Placebo Comparator): no medication before surgery
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: anastrozole — anastrozole 1mg/day 11 days before their surgery and to take the last dose of the oral endocrine agent (anastrozole) on the day before their surgery.
  Arms: 1
Other: Placebo — No medication before surgery
  Arms: 2

SUMMARY:
The purpose of this pilot study is to see if taking anastrozole (Arimidex) for 10 days causes changes in breast cancer cells. Anastrozole (Arimidex) is a drug used in the treatment of a type of breast cancer that depends on estrogen to grow. This type of breast cancer is called estrogen receptor positive breast cancer. Anastrozole (Arimidex) works by blocking an enzyme in your body called aromatase. Aromatase is found in your muscles, fat, liver and in breast tumors. This enzyme is important for making estrogen in women who are no longer having menstrual periods. Anastrozole decreases levels of estrogen in the body. We are interested in seeing if taking anastrozole for 10 days will cause changes in breast cancer cells. We will study cell processes such as how they make new blood vessels, how quickly the cells multiply, and how soon they die. We will also study which genes in the breast cancer tissues are turned on or off by taking anastrozole for 10 days.

DETAILED DESCRIPTION:
This is an exploratory study utilizing micro-array technology and immunohistochemistry to test the hypothesis that changes in gene expression occur as an early event in response to endocrine therapy and that these changes can be correlated with changes in surrogate biological markers.

ELIGIBILITY:
Inclusion Criteria:

* Postmenopausal patients, defined as one or more of the following criteria:

Documented history of bilateral oophorectomy, Aged 60 years or more,

Aged 45-59 years and satisfying one or more of the following criteria:

Amenorrhea for at least 12 months and intact uterus Amenorrhea for less than 12 months and follicle stimulating hormone (FSH) concentrations within postmenopausal range including: patients who have had a hysterectomy and patients who have received hormone replacement therapy in the past.

* Clinically palpable or non-palpable T1c or greater, ER positive invasive breast cancer diagnosed by outside core biopsy.
* Outside diagnosis of invasive breast cancer confirmed at MSKCC
* Palpable or non-palpable breast mass > 1cm highly suspicious for invasive breast cancer based on mammographic, ultrasound and/or physical examination findings and amenable to diagnostic core biopsy.
* Core biopsy diagnosis of ER positive invasive breast cancer performed at MSKCC
* Breast conserving surgery or mastectomy scheduled at MSKCC.
* Informed consent obtained.

Exclusion Criteria:

* Co-morbid conditions which would preclude use of aromatase inhibitors such as: previous hypersensitivity, severe hepatic insufficiency (SGOT or SGPT three times the upper limit of normal), severe renal insufficiency (creatinine clearance <10ml/min).

Prior radiation therapy to chest wall / breast.

* Neoadjuvant chemotherapy
* Hormone replacement therapy, tamoxifen or raloxifene treatment within past 3 months
* ER negative breast cancer
* History of active malignancy within the previous 5 years (except for nonmelanoma skin cancer and breast cancer)

Min Age: 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2004-03; Primary Completion 2009-11 (Actual); Study Completion 2009-11 (Actual)

PRIMARY OUTCOMES:
To determine whether short term exposure to endocrine therapy (anastrozole) induces changes in gene expression in human invasive breast cancer. | conclusion of study

SECONDARY OUTCOMES:
To evaluate the effects of anastrozole-mediated aromatase inhibition on surrogate biomarkers for cell proliferation, apoptosis, and angiogenesis. | conclusion of study

CONTACTS AND LOCATIONS:
Overall Officials: Tari King, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan-Kettering Cancer Center, New York, New York, United States

REFERENCES:
- See also: Memorial Sloan-Kettering Cancer Center — http://www.mskcc.org